CLINICAL TRIAL: NCT06746532
Title: Neonatal Intranasal Breast Milk, Impact on Brain Growth in Hypoxic-ischemic Encephalopathy Therapy (NEO-BRIGHT)
Brief Title: Intranasal Breast Milk Therapy in HIE
Acronym: NEO-BRIGHT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNGYK/40202-5/2024
Record Dates: First submitted 2024-12-16; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Hypoxic-Ischaemic Encephalopathy; Neonatal Encephalopathy; Perinatal Asphyxia; Neonatal Hypoxic Ischemic Encephalopathy
Keywords: HIE; intranasal breast milk; perinatal asphyxia; brain; breast milk stem cells; hypoxic-ischemic encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard care for moderate or severe hypoxic-ischemic encephalopathy with hypothermia.
- Intranasal breast milk (Experimental): Fresh own mother's breast milk expressed within 4 hours, will be administered 2 times daily, 0.4 ml in each nostril for 28 days.
  Interventions: Biological: Intranasal breast milk

INTERVENTIONS:
Biological: Intranasal breast milk — Own-mother's fresh breast milk (within 4 hours of having been expressed), is administered intranasally to neonates with hypoxic-ischemic encephalopathy receiving therapeutic hypothermia, starting from the first day of life and continuing for 28 days.
  Dose: 2 times daily, 0.4 ml in each nostril.
  Arms: Intranasal breast milk

SUMMARY:
This is an open-label prospective single-center randomized controlled trial to evaluate the effect of intranasal breast milk in hypoxic-ischemic encephalopathic neonates receiving therapeutic hypothermia on long term neurodevelopmental outcome compared to standard care.

DETAILED DESCRIPTION:
Perinatal asphyxia and the resulting hypoxic-ischemic encephalopathy (HIE) are the leading cause of neonatal mortality and long-term neurodevelopmental disabilities. Based on our current knowledge, therapeutic hypothermia is the only therapy that has been proven to reduce central nervous system damage in HIE neonates. Improving neurodevelopmental outcomes of newborns with HIE has been an intense area of research over the past decade.

Breast milk is a complex biological substance that contains a variety of bioactive components including neurotrophic growth factors, cytokines, immunoglobulins, and multipotent stem cells. Studies have shown that exclusive breastfeeding in the early stages of development has a positive impact on cognitive outcomes. Animal studies support that mesenchymal stem cells and neurotrophic substances found in breast milk, when administered intranasally enter the central nervous system and reduce the extent of neurological damage. In preterm infants, it has been shown that intranasally administered breast milk is safe and well-tolerated.

In this open-label prospective randomized controlled single-center interventional study, the objective is to administer fresh, own-mother's breast milk intranasally to neonates with hypoxic-ischemic encephalopathy receiving therapeutic hypothermia, starting from the first day of life and continuing for 28 days.

The primary objective is to compare neurodevelopmental outcomes between the control group and the intervention group receiving intranasal breast milk treatment. The secondary objective is to compare the progression of enteral feeding and the duration of exclusive breastfeeding between the intervention and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe hypoxic- ischemic encephalopathy, receiving therapeutic hypothermia

  ≥ 35. gestational week < 48 hours of life
* Hypothermia treatment for 72 hours
* Parental consent form

Exclusion Criteria:

* Congenital malformation
* Concurrent cerebral lesions
* ECMO therapy
* Contraindication of lactation
* Mother unable or unwilling to provide fresh breast milk
* Postpartum asphyxia

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental outcome | 2 years
  The primary outcome will be the 2 year neurodevelopmental outcome comparing standard care and intranasal breast milk therapy groups.
  The Bayley Scales of Infant Development, Third Edition (Bayley-III) score will be used to assess neurodevelopmental outcome, favorable outcome is defined as having composite scores for cognitive, language and motor scales >85, while adverse outcome is defined as composite scores <80 or death.

SECONDARY OUTCOMES:
Time to reach full enteral feeding | 1 month
  Time to reach full enteral feeding will be recorded and analyzed as a secondary outcome.
Length of exclusive breast feeding | 2 years
  Lengths of exclusive breast feeding will be recorded and analyzed as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Unoke Meder, MD, PhD, Principal Investigator — Department of Neonatology, Pediatric Center, Semmelweis University, Budapest, Hungary
Locations (1):
- Department of Neonatology, Pediatric Center, Semmelweis University, Budapest, Hungary, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
On special request pending data transfer agreement approval by Semmelweis University.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 20.12.2024.-01.01.2030.
Access Criteria: On special request pending data transfer agreement approval by Semmelweis University. Sharing upon reasonable request.
URL: https://semmelweis.hu/bokayklinika/kutatas/asphyxia-munkacsoport/

REFERENCES:
- [Background] Chen Y, Zhang C, Huang Y, Ma Y, Song Q, Chen H, Jiang G, Gao X. Intranasal drug delivery: The interaction between nanoparticles and the nose-to-brain pathway. Adv Drug Deliv Rev. 2024 Apr;207:115196. doi: 10.1016/j.addr.2024.115196. Epub 2024 Feb 7. PMID 38336090
- [Background] Baak LM, Wagenaar N, van der Aa NE, Groenendaal F, Dudink J, Tataranno ML, Mahamuud U, Verhage CH, Eijsermans RMJC, Smit LS, Jellema RK, de Haan TR, Ter Horst HJ, de Boode WP, Steggerda SJ, Prins HJ, de Haar CG, de Vries LS, van Bel F, Heijnen CJ, Nijboer CH, Benders MJNL. Feasibility and safety of intranasally administered mesenchymal stromal cells after perinatal arterial ischaemic stroke in the Netherlands (PASSIoN): a first-in-human, open-label intervention study. Lancet Neurol. 2022 Jun;21(6):528-536. doi: 10.1016/S1474-4422(22)00117-X. PMID 35568047
- [Background] Hoban R, Gallipoli A, Signorile M, Mander P, Gauthier-Fisher A, Librach C, Wilson D, Unger S. Feasibility of intranasal human milk as stem cell therapy in preterm infants with intraventricular hemorrhage. J Perinatol. 2024 Nov;44(11):1652-1657. doi: 10.1038/s41372-024-01982-8. Epub 2024 Apr 30. PMID 38688998
- [Background] Keller T, Korber F, Oberthuer A, Schafmeyer L, Mehler K, Kuhr K, Kribs A. Intranasal breast milk for premature infants with severe intraventricular hemorrhage-an observation. Eur J Pediatr. 2019 Feb;178(2):199-206. doi: 10.1007/s00431-018-3279-7. Epub 2018 Nov 1. PMID 30386923